CLINICAL TRIAL: NCT03673709
Title: Group Antenatal Care: Effectiveness for Maternal/Infant and HIV Prevention Outcomes and Contextual Factors Linked to Implementation Success in Malawi
Brief Title: Group Antenatal Care: Effectiveness and Contextual Factors Linked to Implementation Success in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Malawi (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Crystal L. Patil, PhD, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-0845; R01NR018115 (NIH)
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Prenatal Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research team working on the effectiveness evaluation of group care is blinded to study condition and is charged with collecting the Aim 1 effectiveness data from the individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Antenatal Care (usual care) (No Intervention): Women are provided antenatal care services on a first come, first serve basis and listen to a health lecture. They meet individually with a midwife for a physical assessment. Women complete laboratory tests (including HIV testing) at their first visit. Congruent with the new WHO recommendations, individual antenatal care consists of 8 antenatal care visits and 2 postnatal visits at 1 week and 6 weeks.
- Group Antenatal Care (intervention) (Experimental): Women have the same number of visits as those in individual care. Their first antenatal care (intake) and first postnatal visit is done individually (identical to individual care). Women in group care bypass the waiting area and have a 2-hour visit with the same provider in a group of 8-12 women at a similar stage of pregnancy. Women assess their blood pressure and weight, briefly consult the midwife in a corner of the room, and meet for 80-90 minutes of interactive health promotion, enlivened by games and role-plays.
  Interventions: Behavioral: Antenatal Care

INTERVENTIONS:
Behavioral: Antenatal Care — Women in group care bypass the waiting room and have a 2-hour visit with the same provider with a group of 8-12 women at a similar stage of pregnancy. Women assess their own blood pressure and weight, briefly consult the midwife in a corner of the room, and meet for 80-90 minutes of interactive health promotion, enlivened by games and role-plays.
  Arms: Group Antenatal Care (intervention)

SUMMARY:
In this study, we test the effectiveness of an evidence-based model of group antenatal care by comparing it to individual (usual) antenatal care. We simultaneously identify the degree of implementation success and the contextual factors associated with success across 6 antenatal clinics in Blantyre District, Malawi. If results are negative, governments will avoid spending on ineffective care. Positive maternal, neonatal and HIV-related outcomes of group antenatal care will save lives, impact the cost and quality of antenatal care, and influence health policy as governments adopt this innovative model of care nationally.

DETAILED DESCRIPTION:
Sub-Saharan Africa has the world's highest rates of maternal and perinatal mortality and accounts for 2/3 of new HIV infections and 1/4 of preterm births. Antenatal (prenatal) care is the entry point into the health system for many women and offers a unique opportunity to provide life-saving monitoring. However, provider shortages, low quality of care and failure to attend all recommended visits mean that the potential benefits of antenatal care are not realized. There is an urgent need to test novel interventions to reduce health risks for mother and child. Group antenatal care is a transformative model of care that provides a positive pregnancy experience, uses provider time efficiently, and improves perinatal and HIV-related outcomes. Women in group antenatal care have 2-hour visits with the same provider in a group of 8-12 women at a similar stage of pregnancy. Women conduct self-assessments, briefly consult the midwife, and meet for 80-90 minutes of interactive health promotion enlivened by games and role-plays. Women form relationships with midwives and each other. In a US randomized clinical trial (RCT), group care improved prematurity rates, antenatal care attendance, satisfaction with care, breastfeeding practices, safer sex behaviors, and uptake of family planning. Our randomized pilot in Malawi and Tanzania had promising outcomes. More women in group care than in usual care completed ≥4 antenatal visits (94% vs 58%). Their partners were more likely to be tested for HIV during pregnancy (51% vs. 27%). We established that group antenatal care can be offered in a rigorous RCT with high fidelity despite provider shortages. The next step is an adequately powered effectiveness trial. Malawi is an especially appropriate site because it has the world's highest prematurity rate (18%) and high HIV prevalence (10% nationally, 16% at the study site). We use a hybrid design to simultaneously conduct an effectiveness RCT with individual-level randomization and examine implementation processes at 6 clinics in Blantyre District, Malawi. Aim 1 is to evaluate the effectiveness of group antenatal care through 6 months postpartum. We hypothesize that compared to usual care, women in group care and their infants will have less morbidity and mortality and more positive HIV prevention outcomes. We test Aim 1 hypotheses using multi-level hierarchical models using data from repeated surveys and health records. Aim 2 is to identify clinic-level degree of implementation success and contextual factors associated with success for each clinic and across clinics. Analyses use within and across-case matrices. This high-impact study addresses three global health priorities, maternal and infant mortality and HIV prevention, that affect all women of childbearing age in Malawi. The Ministry of Health strongly supports this project; results will help them decide whether to scale-up this innovative model of group care. Negative results will avoid spending on ineffective care. Positive results will provide evidence needed to adopt group antenatal care nationally and in other low-resource countries.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, 24 weeks gestation or less, no marked cognitive impairment, speaks and understands Chichewa (the national language)

Exclusion Criteria:

* Not pregnant, more than 24 weeks gestation, marked cognitive impairment, does not speak or understand Chichewa (the national language)

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1887 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Preterm birth | 8 weeks postpartum
  Newborn born early
Partner HIV Test | Enrollment, 36-42 weeks gestation
  Proportion of partners tested during this pregnancy

SECONDARY OUTCOMES:
Spontaneous abortion | 36-42 weeks gestation
  Pregnancy loss less than 20 weeks
Stillbirth | 8 weeks postpartum
  Baby born with no signs of life at or after 28 weeks gestational age
Low birthweight | 8 weeks postpartum
  Newborn weighing less than 2.5 kg or 2500 grams, measured within 24 hours of birth
Neonatal death | 8 weeks postpartum
  Newborn dies between 0-28 days after birth
Maternal death | 8 weeks postpartum, 6 months postpartum
  Woman dies in pregnancy or within 42 days of the end of pregnancy
Woman HIV test | Enrollment, 36-42 weeks gestation
  Initial HIV test, if seronegative then repeated in 3rd trimester of pregnancy
Anemia | Enrollment, 36-42 weeks gestation; 8 weeks postpartum, 6 months postpartum
  Hemoglobin
Family planning | 8 weeks postpartum; 6 months postpartum
  Using a family planning method (yes/no)
Exclusive breastfeeding | 8 weeks postpartum; 6 months postpartum
  Duration in days
Early repeat pregnancy | 8 weeks postpartum; 6 months postpartum
  Negative pregnancy test and no reported pregnancy loss
ART medication (woman) | Enrollment, 36-42 weeks gestation; 8 weeks postpartum, 6 months postpartum
  Received medication from intake through six months postpartum
HIV test infant | Enrollment, 36-42 weeks gestation; 8 weeks postpartum, 6 months postpartum
  Infant tested for HIV and results received
Self Reporting Questionnaire (SRQ) | Enrollment, 36-42 weeks gestation; 8 weeks postpartum, 6 months postpartum
  The Self Reporting Questionnaire (SRQ) is a brief measure of psychiatric symptomatology designed by the WHO to be used to screen for common mental disorders. It consists of 20 questions with yes/no answers exploring symptoms of depression, anxiety, and somatic complaints such as headache and non-specific gastrointestinal symptoms. SRQ has been translated and validated in several African countries. A recent study conducted in Rwanda reported the α = 0.85 for refugee women. It consists of 20 Yes/No Items, with a total score range from 0-20; α = 0.789. Higher scores indicate more distress.
Satisfaction with care | 36-42 weeks gestation
  10-item satisfaction with antenatal care index; 5 point Likert scale [1 (poor) and to 5 (excellent)], range 10-50, α =0.980
Healthcare utilization | 36-42 weeks gestation; 8 weeks postpartum
  Pre- and postnatal care attendance; health facility birth (yes/no), services received (21 items); content covered (18 items)
Adequate HIV knowledge | Enrollment, 36-42 weeks gestation
  Total HIV Knowledge is the number of questions answered correctly for five HIV-prevention items defined by UNAIDS as essential plus an additional four items from the Malawi Demographic and Health Survey assessing prevention of maternal-to-child transmission. Higher scores indicate more knowledge about how HIV is transmitted.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Patil, PhD, Principal Investigator — University of Illinois at Chicago
Locations (6):
- Malawi (6):
  - Bangwe HC, Blantyre
  - Chileka HC, Blantyre
  - Chilomoni HC, Blantyre
  - Limbe HC, Blantyre
  - Lirangwe HC, Blantyre
  - Madziabango HC, Blantyre

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available to other researchers for secondary analyses after the primary outcome publications have been accepted for publication, approximately 3 years after the grant ends.

REFERENCES:
- [Derived] Patil CL, Norr KF, Kapito E, Liu LC, Mei X, Chodzaza E, Chorwe-Sungani G, Kafulafula U, Abrams ET, Desloge A, Gresh A, Jeremiah RD, Patel DR, Batchelder A, Wang H, Faydenko J, Rising SS, Chirwa E. Group antenatal care positively transforms the care experience: Results of an effectiveness trial in Malawi. PLoS One. 2025 Jun 18;20(6):e0317171. doi: 10.1371/journal.pone.0317171. eCollection 2025. PMID 40531963
- [Derived] Liese KL, Kapito E, Chirwa E, Liu L, Mei X, Norr KF, Patil CL. Impact of group prenatal care on key prenatal services and educational topics in Malawi and Tanzania. Int J Gynaecol Obstet. 2021 Apr;153(1):154-159. doi: 10.1002/ijgo.13432. Epub 2020 Dec 2. PMID 33098114
- [Derived] Chirwa E, Kapito E, Jere DL, Kafulafula U, Chodzaza E, Chorwe-Sungani G, Gresh A, Liu L, Abrams ET, Klima CS, McCreary LL, Norr KF, Patil CL. An effectiveness-implementation hybrid type 1 trial assessing the impact of group versus individual antenatal care on maternal and infant outcomes in Malawi. BMC Public Health. 2020 Feb 10;20(1):205. doi: 10.1186/s12889-020-8276-x. PMID 32039721